CLINICAL TRIAL: NCT07334483
Title: A Randomized, Active-Controlled, Open-Label Study of Yttrium [90Y] Microsphere Injection in Combination With Camrelizumab and/or Apatinib and Yttrium [90Y] Microsphere Injection Alone Versus cTACE in the Treatment of HCC
Brief Title: A Study of Yttrium [90Y] Microsphere Injection in Combination With Targeted Immunotherapy in the Treatment of HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GrandPharma (China) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST561-1
Record Dates: First submitted 2025-08-13; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: HCC
Keywords: Yttrium [90Y] Microsphere Injection
MeSH Terms: interventions — Yttrium; Yttrium-90; Microspheres; camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Yttrium [90Y] microsphere injection selective internal radiation therapy (SIRT) + camrelizumab + apatinib
  Interventions: Drug: Yttrium [90Y] Microsphere Injection; Drug: Camrelizumab; Drug: Apatinib
- Group B (Experimental): Yttrium [90Y] microsphere injection SIRT + camrelizumab
  Interventions: Drug: Yttrium [90Y] Microsphere Injection; Drug: Camrelizumab
- Group C (Experimental): Yttrium [90Y] microsphere injection SIRT
  Interventions: Drug: Yttrium [90Y] Microsphere Injection
- Group D (Active Comparator): Conventional transcatheter arterial chemoembolization
  Interventions: Other: Conventional transcatheter arterial chemoembolization

INTERVENTIONS:
Drug: Yttrium [90Y] Microsphere Injection — Yttrium [90Y] microsphere injection should be implanted through the hepatic artery based on 99mTc-MAA SPECT/CT simulated surgery (Mapping) to evaluate the distribution of microsphere in the body, and calculate the activity required for treatment
  Other Names: Yttrium-90 resin microsphere
  Arms: Group A; Group B; Group C
Other: Conventional transcatheter arterial chemoembolization — For the operation method of cTACE, please refer to the Clinical Practice Guidelines for Transcatheter Arterial Chemoembolization (TACE) Treatment of Hepatocellular Carcinoma in China (2023 Edition) and its related standard operating procedures (SOPs).
  Other Names: cTACE
  Arms: Group D
Drug: Camrelizumab — The first dose of Cycle 1 should be completed within 3 days after randomization. After Cycle 1 Day 1 (C1D1), it should be dosed every 3 weeks ± 3 days. Dosing may be delayed due to holidays, but should not exceed 7 days
  Other Names: CAM
  Arms: Group A; Group B
Drug: Apatinib — Apatinib will be used from Cycle 2 Day 1 (C2D1). Apatinib should be discontinued for at least 7 days before and after treatment with yttrium [90Y] microsphere injection
  Other Names: RIVO
  Arms: Group A

SUMMARY:
This study is A Randomized, Active-Controlled, Open-Label National Multicenter Phase 2 Registration Clinical Study of Yttrium [90Y] Microsphere Injection in Combination with Camrelizumab and/or Apatinib and Yttrium [90Y] Microsphere Injection Alone versus Conventional Transcatheter Arterial Chemoembolization (cTACE) in the Treatment of Unresectable or Non-Ablative, Non-Metastatic Hepatocellular Carcinoma (HCC). Its aim is to evaluate the efficacy and safety of yttrium [90Y] resin microsphere injection combined with Camrelizumab and/or apatinib compared with yttrium [90Y] resin microsphere injection alone in the treatment of inoperable or ablatable, non-metastatic HCC.

DETAILED DESCRIPTION:
This is a prospective, randomized, active-controlled, open-label, multicenter Phase 2 clinical study to evaluate the efficacy and safety of yttrium [90Y] microsphere injection in combination with camrelizumab and/or apatinib and yttrium [90Y] microsphere injection alone versus cTACE in the treatment of unresectable or non-ablative, non-metastatic HCC.

A total of at least 120 subjects with unresectable or non-ablative, non-metastatic HCC are planned to be enrolled and randomly assigned to groups A, B, C and D in a 1:1:1:1 ratio, that is, yttrium [90Y] microsphere injection + camrelizumab + apatinib group (A), yttrium [90Y] microsphere injection + camrelizumab group (B), yttrium [90Y] microsphere injection group (C) and cTACE group (D). The above treatment will continue until the criteria for withdrawal from study treatment are met, whichever occurs first. Subjects will receive yttrium [90Y] microsphere injection alone or in combination with camrelizumab and/or apatinib for up to 18 months.

The primary endpoint of the Phase 2 study is ORR assessed by BICR based on mRECIST criteria. The key secondary endpoint is PFS assessed by BICR based on mRECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily participate in this study, sign the informed consent form (ICF), and are able to comply with the diagnosis, treatment, observation, follow-up visit and related procedures specified in this protocol, with good compliance.
2. Patients aged ≥ 18 and ≤ 75, regardless of gender.
3. HCC confirmed by pathological histology/cytology, or meeting the clinical diagnostic criteria in the Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2024 Edition) established by the National Health Commission.
4. Patients who are not suitable for surgery (including hepatectomy and liver transplantation) or ablation treatment based on the judgment of investigator or clinical practice guidelines, or refuse surgery or ablation treatment.
5. China Liver Cancer Clinical Staging (CNLC): Ib-IIIa. Vp4 portal vein tumor thrombus invasion will be excluded, if combined with Vp1-3 portal vein tumor thrombus, the tumor thrombus must be located on the same side of the liver lobe as the targeted tumor area.
6. Patients with at least 1 measurable lesion according to RECIST v1.1 and mRECIST criteria.
7. Patients who have been evaluated by Yttrium [90Y] Microsphere Injection Selective Internal Radiation Therapy and Dose Evaluation Committee as suitable for SIRT treatment.
8. For yttrium [90Y] microsphere injection, camrelizumab and apatinib, there are no contraindications for use in the product instructions and clinical practice guidelines. Patients who are suitable for cTACE treatment, have no contraindications to use in clinical practice guidelines, are expected to be able to use up to 4 cTACE treatments for localized liver lesions within 24 weeks during the study period, and are expected to receive 1-2 cTACE treatments for a single lesion.
9. ECOG PS score: 0-1.
10. Child-Pugh liver function classification: Class A or Class B with ≤7 points.
11. Life expectancy ≥3 months.
12. If the subject has HBV or HCV infection, the following criteria must be met:

    i. Subjects with HBV infection (HBsAg and/or HBV-DNA positive): Subjects should receive antiviral treatment with one of the 4 drugs recommended by the national clinical guidelines for hepatitis B (tenofovir disoproxil fumarate, tenofovir alafenamide fumarate, tenofovir amibufenamide and entecavir) for at least 7 days before the first study treatment to achieve HBV-DNA < 2000 IU/mL or < 104 copies/mL. The standardized antiviral treatment must be received throughout the study.

    ii. If HCV-Ab is positive, the blood HCV RNA must be negative.
13. Patients who have basically normal organ and bone marrow functions:

    i. Hematology (corrective treatment such as any blood components or cell growth factors is not allowed within 7 days before the laboratory tests): Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelet count (PLT) ≥ 75 × 109/L; hemoglobin (HGB) ≥ 90 g/L.

    ii. Liver function (human albumin or plasma transfusion is not allowed within 7 days before the laboratory tests): Serum total bilirubin (TBIL) ≤ 2 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN, alkaline phosphatase (ALP) ≤ 5 × ULN; serum albumin ≥ 30 g/L.

    iii. Renal function: Serum creatinine (Cr) ≤ 1.5 × ULN, or the calculated value of creatinine clearance (CrCI, estimated according to Cockcroft-Gault formula) ≥ 50 mL/min. Urinalysis results show that urine protein is < 2+ (if urine protein is ≥ 2+, the 24-hour urine protein quantitative test should be performed, and patients can be enrolled if the 24-hour urine protein quantification is < 1.0 g).

    iv. Coagulation function: International normalized ratio (INR) ≤ 1.8, or prothrombin time (PT) exceeds the range of normal control ≤ 4 seconds.
14. Patients of childbearing potential should use effective contraceptive measures from the signing of the ICF to at least 3 months after the last study treatment.

Exclusion Criteria:

1. Cholangiocarcinoma, combined hepatocellular-cholangiocarcinoma, sarcomatoid hepatocellular carcinoma and fibrolamellar hepatocellular carcinoma confirmed by pathological histology or cytology.
2. Invasive HCC, that is, imaging shows that microscopic or small tumor nodules are diffusely distributed in a certain liver lobe or the entire liver.
3. Based on liver volume, the tumor burden is relatively large (>50%).
4. Presence of hepatic vein or inferior vena cava tumor thrombus, or involvement of the superior mesenteric vein or more distant end.
5. Patients with other malignant tumors other than HCC within 5 years or at the same time. However, patients with cured localized tumors such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate cancer in situ, cervical cancer in situ and breast cancer in situ can be enrolled.
6. Conversion therapies such as interventional and targeted immunotherapy have been used before hepatectomy, including conversion of functional residual liver volume (using ALPPS or PVE) and oncology conversion therapy.
7. Previous systemic anti-tumor treatment for HCC, including molecular targeted drugs, systemic chemotherapy and immunotherapy (immune checkpoint inhibitors, antibody-drug conjugate [ADC], immune cells, oncolytic viruses and tumor vaccines, etc.).
8. Use of Chinese patent medicines and modern Chinese medicine preparations with anti-liver cancer indications within 7 days before randomization.
9. Previous local treatment for liver lesions, including TACE, transarterial embolization (TAE), hepatic artery infusion chemotherapy (HAIC), radiotherapy, or ablation of target liver lesions, injection of oncolytic viruses, and internal/external radiation therapy. In the case of adjuvant therapy after radical resection, patients who have only received one TACE can be enrolled.
10. Previous solid organ (such as liver transplantation) or allogeneic stem cell transplantation (except for patients who have only received corneal transplantation).
11. Patients with bile duct obstruction due to any reason that has not been resolved before randomization.
12. Patients with decompensated cirrhosis and severe liver function impairment (Child-Pugh Grade C) before randomization, including severe jaundice, hepatic encephalopathy, hepatorenal syndrome or refractory ascites (i.e. clinically symptomatic moderate or severe ascites requiring therapeutic puncture, drainage or Child-Pugh ascites score > 2).
13. Patients with clinically symptomatic pleural effusion and pericardial effusion requiring puncture and drainage before randomization. However, patients who have received puncture and drainage within 2 weeks before enrollment and only show a small amount of effusion on imaging without clinical symptoms can be enrolled.
14. History of iodine contrast agent allergy of grade II or above, or inability to undergo enhanced liver CT scan due to any reason.
15. Patients who are unable to swallow the drug, have malabsorption syndrome, incomplete gastrointestinal obstruction or any condition that significantly affects the gastrointestinal absorption of apatinib mesylate before randomization.
16. History of active pulmonary tuberculosis. For subjects suspected of having active pulmonary tuberculosis, the definitive diagnosis should be made in combination with chest imaging, sputum, clinical symptoms and signs.
17. Patients with congenital or acquired immune deficiency (such as HIV infection), active syphilis, or co-infection of hepatitis B and C.
18. Patients with clinically significant cardiovascular and cerebrovascular diseases before randomization:

    i. Uncontrollable hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) after optimal antihypertensive treatment, with a previous history of hypertensive crisis or hypertensive encephalopathy.

    ii. History of myocardial infarction, unstable angina pectoris, cerebral infarction, cerebral haemorrhage or any other major cardiovascular and cerebrovascular accident within 6 months before randomization.

    iii. Congestive heart failure classified as grade 2 or above by the New York Heart Association (NYHA): Left ventricular ejection fraction (LVEF) < 50%.

    iv. Severe cardiac rhythm or conduction abnormalities, including supraventricular or ventricular arrhythmias requiring treatment, QTcF value ≥ 450 ms (males)/≥ 470 ms (females), or second-degree or third-degree atrioventricular block.

    v. History of myocarditis or related examinations suggest active myocarditis. vi. Subjects with heart disease who are assessed by the investigator to be intolerant of other tests.
19. Patients with a history of interstitial pneumonia or interstitial lung disease, or a previous history of interstitial pneumonia or interstitial lung disease requiring corticosteroid therapy, or other pulmonary fibrosis and organising pneumonia that may interfere with the judgment and treatment of immune/SIRT-related pulmonary toxicity.
20. Patients with severe hemorrhagic tendency or coagulation dysfunction, or receiving thrombolytic therapy; patients who have received or are receiving conventional doses of nonsteroidal anti-inflammatory drugs (such as aspirin, indomethacin ibuprofen and naproxen), antiplatelet drugs (such as clopidogrel, ticlopidine, dipyridamole and cilostazol) or anticoagulants (such as warfarin and low molecular weight heparin) within 10 days before randomization.
21. Subjects who have participated in other clinical studies and used the investigational drug or device within 30 days before randomization.
22. Patients with active autoimmune diseases requiring systemic treatment (such as the use of disease-modifying drugs, corticosteroids or immunosuppressive agents) within 1 year before randomization or a history of autoimmune diseases that may recur. Patients receiving replacement therapy (such as thyroid hormone replacement therapy for hypothyroidism, type 1 diabetes mellitus requiring only insulin replacement therapy, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) can be enrolled.
23. Subjects at risk of bleeding, as follows:

    i. Subjects with history of gastrointestinal bleeding or a significant tendency to gastrointestinal bleeding within 6 months before randomization, such as esophageal or gastric variceal bleeding caused by portal hypertension, local active peptic ulcer or persistent faecal occult blood positive.

    ii. Any life-threatening bleeding event within 3 months before randomization, including the events requiring blood transfusion, surgery or local treatment, and continuous drug therapy.

    iii. Subjects with esophageal or gastric varices requiring interventional treatment within 28 days before randomization.

    iv. Untreated or incompletely treated esophageal or gastric fundus varices that are at high risk of bleeding as judged by the investigator.
24. Abdominal fistula, gastrointestinal perforation or abdominal abscess within 6 months before randomization.
25. Patients with intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction within 6 months before randomization, including incomplete obstruction related to pre-existing diseases or requiring routine parenteral hydration, parenteral nutrition or tube feeding.
26. History of deep vein thrombosis, pulmonary embolism or any other serious thromboembolism within 3 months before randomization (except for implantable venous access port or catheter-related thrombosis, or superficial vein thrombosis).
27. Patients who have undergone major surgery or serious trauma within 28 days before randomization (and cannot participate in the study as judged by the investigator); patients with severe unhealed wound, active ulcer or untreated fracture before randomization.
28. Patients who have received live attenuated vaccine or treatment within 28 days before randomization.
29. Use of strong CYP3A4 inducers or strong CYP3A4 inhibitors within 7 days before randomization.
30. Use of immunosuppressive agents or systemic corticosteroids therapy for immunosuppression within 14 days before randomization, excluding topical corticosteroids or systemic application of low-dose prednisone (not more than 10 mg/day) or equivalent doses of other corticosteroids.
31. Patients who have received drugs with immunomodulatory effects within 14 days before randomization, including systemic use of thymosin-α1, interferon and interleukin-II.
32. Pregnant or lactating women, or women who need to continue breastfeeding during the study.
33. Any other serious diseases, metabolic disorders or laboratory test abnormalities that are not suitable for treatment with the investigational drug, will affect the interpretation of the study results, or put the patient at high risk as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 18 months
  Objective Response Rate, assessed by blinded independent central review (BICR) based on mRECIST criteria

SECONDARY OUTCOMES:
PFS | up to 18 months
  Progression-free survival (PFS, assessed by BICR based on mRECIST and RECIST v1.1 criteria)
ORR | up to 18 months
  Objective Response Rate (assessed by BICR based on RECIST v1.1 criteria)
hPFS | up to 18 months
  Hepatic Progression-free survival (hPFS) (assessed by BICR and investigator based on mRECIST criteria)
hORR | up to 18 months
  Hepatic Objective Response Rate (hORR) (assessed by BICR and investigator based on mRECIST criteria)
PFS rate | up to 9 months
  Progression-free survival rate at month 9(assessed by BICR based on mRECIST and RECIST v1.1 criteria respectively)
DoR | up to 9 months
  duration of response (DoR)at month 9 (assessed by BICR based on mRECIST and RECIST v1.1 criteria respectively)
DCR | up to 9 months
  Disease control rate (DCR)at month 9 (assessed by BICR based on mRECIST and RECIST v1.1 criteria respectively)
TTP | up to 9 months
  Time to progress (TTP) at month 9 (assessed by BICR based on mRECIST and RECIST v1.1 criteria respectively)
TTR | up to 9 months
  Time to tumor response (TTR)at month 9 (assessed by BICR based on mRECIST and RECIST v1.1 criteria respectively)
OS rate | 12/18/24 months after the first treatment
  Overall survival (OS) rates at months 12/18/24
OS | up to 18 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Zhiping Yan, MD, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Nanjing Tianyinshan Hospital, Nanjin
  - Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No